CLINICAL TRIAL: NCT00522184
Title: Intra-Articular Injection of Etanercept in Patient Suffering From Rheumatoid Arthritis : a Double-Blind Randomized Study for Evaluation of Efficacy and Safety of Etanercept Versus Intra-Articular Steroid Injection in Acute Synovitis
Brief Title: Intra-Articular Injection of Etanercept in Patient Suffering From Rheumatoid Arthritis : a Double-Blind Randomized Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-PP-04
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
Keywords: intra-articular injection; acute synovitis; etanercept
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patient receiving etanercept intra-articular injection
  Interventions: Procedure: intra-articular injection of etanercept
- 2 (Active Comparator): patient receiving steroid intra-articular injection
  Interventions: Procedure: intra-articular injection of steroid

INTERVENTIONS:
Procedure: intra-articular injection of etanercept
  Arms: 1
Procedure: intra-articular injection of steroid
  Arms: 2

SUMMARY:
Intra-articular injection of etanercept in patient suffering from rheumatoid arthritis: a double-blind randomized study for evaluation of efficacy and safety of etanercept versus intra-articular steroid injection in acute synovitis (knee,wrist,ankle,elbow)

ELIGIBILITY:
Inclusion Criteria:

* must be able to understand the information about the study
* diagnosis of rheumatoid arthritis for 6 month at least
* suffering for 2 weeks at least
* with evaluation of pain over 4/10
* with stable DMARDs treatment for three month at least

Exclusion Criteria:

* infection or surgery on the target joint
* treated with infliximab,adalimumab or anakinra

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-02; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Pain | every month during six month

CONTACTS AND LOCATIONS:
Overall Officials: Christian H ROUX, Principal Investigator — Rheumatology department, Nice
Locations (1):
- Rheumatology department, Hopital Archet I, Nice, France